CLINICAL TRIAL: NCT03012594
Title: A Pilot Study to Evaluate Safety and Effectiveness of Lanreotide in the Treatment of Patients With Small Bowel Motility Disorders (SBMD): a Prospective, Non-randomized, Single-center Study of 20 Participants
Brief Title: Lanreotide in the Treatment of Small Bowel Motility Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Ipsen (Industry)
Responsible Party: Principal Investigator, Larry Miller, Chief of Gastroenterology, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS16-0465
Record Dates: First submitted 2017-01-04; First posted 2017-01-06 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Gastrointestinal Motility Disorder; Intestinal Disease
Keywords: Small bowel motility disorder; Slow intestinal motility; Small bowel bacterial overgrowth
MeSH Terms: conditions — Intestinal Diseases | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lanreotide (Experimental): Open label
  Interventions: Drug: Lanreotide

INTERVENTIONS:
Drug: Lanreotide — Dosage: 120mg Dosage form: subcutaneous injection, pre-filled syringe Dosage frequency: 3 injections over 12 weeks, each dose administered 4 weeks apart
  Other Names: Somatuline

SUMMARY:
This is a human research study looking at the effectiveness of Lanreotide (study medication) in treating small bowel motility disorders. It is similar to a natural hormone somatostatin that is produced in the body in the stomach, duodenum, pancreas and brain. Somatostatin is a growth hormone-inhibiting hormone. Lanreotide is a man made hormone and is a long acting medication that is given once a month. It is marketed with a trade name "Somatuline Depot". It is given deep subcutaneously (deep within the layers of the skin) in the superior external quadrant of the buttock. Injection site will be alternated on subsequent injections.

DETAILED DESCRIPTION:
The investigators hypothesize that in patients with small bowel motility disorders, Lanreotide helps in alleviating the symptoms. Lanreotide is an FDA approved medication for management of acromegaly and neuroendocrine tumors, but has never been used for treating small bowel motility disorders. However, Octreotide which is similar to Lanreotide but is a short acting synthetic somatostatin has been used in few research studies.

If a patient is interested and qualifies for the study then he/she will be explained about the study and signature will be collected on the consent form. Health and social history will be collected. Blood work, urine analysis, pregnancy test (in women of reproductive age group and have the capability of getting pregnant)) will be performed to make sure that patient qualifies for the study and for follow-up during the treatment. Physical examination, ECG, wireless motility capsule testing and hydrogen breath testing will be performed. Patients will be required to complete a questionnaire regarding their health.

The total study duration from the first administration of study drug is 12 weeks. The study medication will be given once a month for 3 months and there is a 1 month follow-up after the last study medication. There will be a screening visit approximately 1 month before the first study drug administration.

ELIGIBILITY:
Inclusion Criteria:

1. Consecutive patients with evidence of small bowel motility disorders, referred to (or) are patients of the Gastroenterology and Motility Center at Northwell Health System.
2. Aged between 18 and 70 years.
3. Subjects should be capable of understanding the study and be able to give informed consent.
4. Patient having small bowel motility disorder as evidenced by delayed small bowel transit by wireless motility capsule (WMC) testing to > 6 hours.
5. To participate in the study, patients will have to stop taking Octreotide (because it has the same mechanism of action as the study medication) if they are currently taking it; it should be stopped for at least 4 weeks before taking the first dose of this study medication.

General Exclusion Criteria

1. Age <18 or age >70
2. Pregnancy as assessed by urine pregnancy test.

Exclusion Criteria for performing wireless motility capsule testing

1. History of gastric bezoar
2. History of Disorders of swallowing
3. Known or suspected small bowel diverticula, diverticulitis, strictures, fistulas, Crohn's disease, or any other relevant medical comorbidity (e.g. chronic alcohol abuse)
4. Prior intestinal surgery, including Ileocecal(IC) valve resection or gastrointestinal surgeries that create a blind loop (e.g. Bilroth II or Roux-en-Y)
5. History of Severe dysphagia to food or pills
6. A participant who uses an implanted or portable electro-mechanical medical device such as a cardiac pacemaker or infusion pump
7. Inability to be off intestinal transit altering medication for at least one week (e.g. opiates, laxatives, etc.)
8. Any person unable or unwilling to undergo abdominal surgery.
9. BMI > 40.

Exclusion Criteria due to Lanreotide

1. Current use or recent (within last 7 days) use of acid suppressive therapy, prokinetic agents, laxatives, and opiates, or other agents known to affect gastrointestinal motility.
2. Disorders associated with presumed small intestinal motility disorders including: scleroderma, intestinal pseudo-obstruction, and autonomic visceral neuropathy (e.g. longstanding diabetes of more than 20 years and/or poorly controlled diabetes (glucose > 250, glycosylated hemoglobin (HbA1c) > 8.5%)
3. Current use of cyclosporine (Gengraf, Neoral, or Sandimmune), a medicine called bromocriptine (Parlodel, Cycloset), or medicines that lower heart rate, such as beta blockers.
4. Cardiac arrhythmia based on health history (palpitations, feeling a pause between heartbeats, lightheadedness, passing out, shortness of breath, or chest pain).

   Bradycardia and Tachycardia are monitored during every visit to the clinic, using pulse rate.

   ECG will be performed during screening visit and during 8th week of the study. The following are accessed with ECG.
   * Bradycardia <60 beats/min.
   * Tachycardia >100 beats/min.
   * Atrial Fibrillation - Rapid irregular atrial signal with no real P-waves and irregular ventricular rate.
   * Ventricular Fibrillation - Irregular ventricular waveforms.
   * Sinus Arrhythmia - Normal beats, but triggered at an irregular interval from 60 to 100 beats per minute, causing varying R-R interval.
   * Missed beats.
5. Chronic kidney disease (moderate and severe renal impairment as calculated by creatinine clearance of <50 mL/min)
6. Hepatic Impairment - Subjects with Child-Pugh Class B and Class C.
7. Significant electrolyte abnormalities: Anything outside of the normal range by +/- 20 % will be considered as abnormal.
8. Cholelithiasis (Total bilirubin >2x of normal)
9. Pancreatitis
10. Hepatitis (Aspartate transaminase (AST), Alanine transaminase (ALT) or Alkaline phosphatase (Alk Ph), greater than upper limit of normal(ULN), Serum albumin <3.0 g/dL unless prothrombin time is within the normal range)
11. Present cholecystitis
12. Uncontrolled congestive heart failure
13. Known hypersensitivity to the study drug

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-11 (Actual); Primary Completion 2018-10-21 (Actual); Study Completion 2019-03-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Miller, M.D., Principal Investigator — Northwell Health
Locations (2):
- United States (2):
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Lenox Hill Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soudah HC, Hasler WL, Owyang C. Effect of octreotide on intestinal motility and bacterial overgrowth in scleroderma. N Engl J Med. 1991 Nov 21;325(21):1461-7. doi: 10.1056/NEJM199111213252102. PMID 1944424
- [Background] Owyang C. Octreotide in gastrointestinal motility disorders. Gut. 1994;35(3 Suppl):S11-4. doi: 10.1136/gut.35.3_suppl.s11. PMID 8206395
- [Background] Edmunds MC, Chen JD, Soykan I, Lin Z, McCallum RW. Effect of octreotide on gastric and small bowel motility in patients with gastroparesis. Aliment Pharmacol Ther. 1998 Feb;12(2):167-74. doi: 10.1046/j.1365-2036.1998.00289.x. PMID 9692691
- [Background] Faure C, Goulet O, Ategbo S, Breton A, Tounian P, Ginies JL, Roquelaure B, Despres C, Scaillon M, Maurage C, Paquot I, Hermier M, De Napoli S, Dabadie A, Huet F, Baudon JJ, Larchet M. Chronic intestinal pseudoobstruction syndrome: clinical analysis, outcome, and prognosis in 105 children. French-Speaking Group of Pediatric Gastroenterology. Dig Dis Sci. 1999 May;44(5):953-9. doi: 10.1023/a:1026656513463. PMID 10235603
- [Background] Stanghellini V, Cogliandro RF, de Giorgio R, Barbara G, Salvioli B, Corinaldesi R. Chronic intestinal pseudo-obstruction: manifestations, natural history and management. Neurogastroenterol Motil. 2007 Jun;19(6):440-52. doi: 10.1111/j.1365-2982.2007.00902.x. PMID 17564625
- [Background] Mann SD, Debinski HS, Kamm MA. Clinical characteristics of chronic idiopathic intestinal pseudo-obstruction in adults. Gut. 1997 Nov;41(5):675-81. doi: 10.1136/gut.41.5.675. PMID 9414977
- [Background] Lybaert W. The use of lanreotide autogel(R) in the treatment of intestinal obstruction in a patient with adenocarcinoma. Case Rep Oncol. 2014 Jan 16;7(1):43-6. doi: 10.1159/000358124. eCollection 2014 Jan. PMID 24575015
- [Background] Lamrani A, Vidon N, Sogni P, Nepveux P, Catus F, Blumberg J, Chaussade S. Effects of lanreotide, a somatostatin analogue, on postprandial gastric functions and biliopancreatic secretions in humans. Br J Clin Pharmacol. 1997 Jan;43(1):65-70. doi: 10.1111/j.1365-2125.1997.tb00034.x. PMID 9056054
- [Background] Camilleri M. Small bowel motility disorders. Rev Gastroenterol Mex. 1994 Apr-Jun;59(2):120-6. PMID 7991964
- [Background] Wang C, Xu H, Chen H, Li J, Zhang B, Tang C, Ghishan FK. Somatostatin stimulates intestinal NHE8 expression via p38 MAPK pathway. Am J Physiol Cell Physiol. 2011 Feb;300(2):C375-82. doi: 10.1152/ajpcell.00421.2010. Epub 2010 Nov 24. PMID 21106692
- [Background] Giustina A, Chanson P, Bronstein MD, Klibanski A, Lamberts S, Casanueva FF, Trainer P, Ghigo E, Ho K, Melmed S; Acromegaly Consensus Group. A consensus on criteria for cure of acromegaly. J Clin Endocrinol Metab. 2010 Jul;95(7):3141-8. doi: 10.1210/jc.2009-2670. Epub 2010 Apr 21. PMID 20410227
- [Background] Wyrwich KW, Mody R, Larsen LM, Lee M, Harnam N, Revicki DA. Validation of the PAGI-SYM and PAGI-QOL among healing and maintenance of erosive esophagitis clinical trial participants. Qual Life Res. 2010 May;19(4):551-64. doi: 10.1007/s11136-010-9620-x. Epub 2010 Feb 27. PMID 20195905
- [Background] Revicki DA, Rentz AM, Tack J, Stanghellini V, Talley NJ, Kahrilas P, De La Loge C, Trudeau E, Dubois D. Responsiveness and interpretation of a symptom severity index specific to upper gastrointestinal disorders. Clin Gastroenterol Hepatol. 2004 Sep;2(9):769-77. doi: 10.1016/s1542-3565(04)00348-9. PMID 15354277
- [Background] Rentz AM, Kahrilas P, Stanghellini V, Tack J, Talley NJ, de la Loge C, Trudeau E, Dubois D, Revicki DA. Development and psychometric evaluation of the patient assessment of upper gastrointestinal symptom severity index (PAGI-SYM) in patients with upper gastrointestinal disorders. Qual Life Res. 2004 Dec;13(10):1737-49. doi: 10.1007/s11136-004-9567-x. PMID 15651544
- [Background] De Giorgio R, Sarnelli G, Corinaldesi R, Stanghellini V. Advances in our understanding of the pathology of chronic intestinal pseudo-obstruction. Gut. 2004 Nov;53(11):1549-52. doi: 10.1136/gut.2004.043968. PMID 15479666
- [Background] Iida H, Ohkubo H, Inamori M, Nakajima A, Sato H. Epidemiology and clinical experience of chronic intestinal pseudo-obstruction in Japan: a nationwide epidemiologic survey. J Epidemiol. 2013;23(4):288-94. doi: 10.2188/jea.je20120173. PMID 23831693
- [Background] Goulet O, Sauvat F, Jan D. Surgery for pediatric patients with chronic intestinal pseudo-obstruction syndrome. J Pediatr Gastroenterol Nutr. 2005 Sep;41 Suppl 1:S66-8. doi: 10.1097/01.scs.0000180312.55417.8e. No abstract available. PMID 16131977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject was enrolled on 5/11/2017 and the last subject was enrolled on 7/19/2018. All study visits were performed either at a medical clinic or gastroenterology unit. There were also phone follow-ups.
Pre-assignment Details: This is an open label non-randomized study. All enrolled participants were checked to see if they meet all the screening requirements to participate. All willing and qualified participants received the study mediation.
Period: Overall Study
Arm/Group | Lanreotide
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Lanreotide
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.78 (13.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 6
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: Participants]
  United States | 9
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.11 (6.8)
Heart rate [Mean (Standard Deviation); unit: beats/sec] | 70.67 (10.91)
Systolic Blood pressure [Mean (Standard Deviation); unit: mmHg] | 120 (19)
Diastolic blood pressure [Mean (Standard Deviation); unit: mmHg] | 77 (8)
Blood Glucose [Mean (Standard Deviation); unit: mg/dL] | 118 (75)
Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index_Heartburn/regurgitation [Mean (Standard Deviation); unit: units on a scale] — The participant rated each of the measured gastrointestinal symptom severity as described below. (Minimum of 0 and a Maximum of 5.) 0=No symptom, 1=Very Mild Symptom, 2= Mild Symptoms, 3= Moderate symptom, 4=Severe symptom, 5= Very Severe symptom.
  This subscale accessed the following 7 symptoms -
  1. Heartburn during day
  2. Regurgitation during day
  3. Heartburn when lying
  4. Regurgitation when lying
  5. Chest discomfort during day
  6. Bitter taste in mouth
  7. Chest discomfort at night
  The computed score is an average of all these gastrointestinal symptoms.
  units on a scale | 1.73 (1.85)
Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index_Nausea/vomiting [Mean (Standard Deviation); unit: units on a scale] — The participant rated each of the measured gastrointestinal symptom severity as described below. (Minimum of 0 and a Maximum of 5.) 0=No symptom, 1=Very Mild Symptom, 2= Mild Symptoms, 3= Moderate symptom, 4=Severe symptom, 5= Very Severe symptom.
  This subscale accessed the following 3 symptoms -
  1. Nausea
  2. Retching
  3. Vomiting
  The computed score is an average of all these gastrointestinal symptoms.
  units on a scale | 1.85 (2.07)
Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index_Fullness/early satiety [Mean (Standard Deviation); unit: units on a scale] — The participant rated each of the measured gastrointestinal symptom severity as described below. (Minimum of 0 and a Maximum of 5.) 0=No symptom, 1=Very Mild Symptom, 2= Mild Symptoms, 3= Moderate symptom, 4=Severe symptom, 5= Very Severe symptom.
  This subscale accessed the following 4 symptoms -
  1. Stomach fullness
  2. Loss of appetite
  3. Not able to finish meal
  4. Excessively full after meal
  The computed score is an average of all these gastrointestinal symptoms.
  units on a scale | 3.22 (1.84)
Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index_Bloating [Mean (Standard Deviation); unit: units on a scale] — The participant rated each of the measured gastrointestinal symptom severity as described below. (Minimum of 0 and a Maximum of 5.) 0=No symptom, 1=Very Mild Symptom, 2= Mild Symptoms, 3= Moderate symptom, 4=Severe symptom, 5= Very Severe symptom.
  This subscale accessed the following 2 symptoms -
  1. Bloating
  2. Stomach visibly larger
  The computed score is an average of all these gastrointestinal symptoms.
  units on a scale | 3.67 (1.57)
Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index_Upper abdominal pain [Mean (Standard Deviation); unit: units on a scale] — The participant rated each of the measured gastrointestinal symptom severity as described below. (Minimum of 0 and a Maximum of 5.) 0=No symptom, 1=Very Mild Symptom, 2= Mild Symptoms, 3= Moderate symptom, 4=Severe symptom, 5= Very Severe symptom.
  This subscale accessed the following 2 symptoms -
  1. Upper abdominal pain
  2. Upper abdominal discomfort
  The computed score is an average of all these gastrointestinal symptoms.
  units on a scale | 2.5 (1.86)
Patient Assessment of Gastrointestinal Disorders-Symptom Severity Index_Lower abdominal pain [Mean (Standard Deviation); unit: units on a scale] — The participant rated each of the measured gastrointestinal symptom severity as described below. (Minimum of 0 and a Maximum of 5.) 0=No symptom, 1=Very Mild Symptom, 2= Mild Symptoms, 3= Moderate symptom, 4=Severe symptom, 5= Very Severe symptom.
  This subscale accessed the following 2 symptoms -
  1. Lower abdominal pain
  2. Lower abdominal discomfort
  The computed score is an average of all these gastrointestinal symptoms.
  units on a scale | 2.83 (1.62)
Gastric emptying time [Mean (Standard Deviation); unit: minutes] | 323 (232)
Small bowel transit time [Mean (Standard Deviation); unit: minutes] | 505 (159)
Colonic transit time [Mean (Standard Deviation); unit: minutes] | 2503 (1592)
Small bowel and colonic transit time [Mean (Standard Deviation); unit: minutes] | 2835 (1556)
Whole gut transit time [Mean (Standard Deviation); unit: minutes] | 3160 (1533)
Stomach Contractions [Mean (Standard Deviation); unit: Contractions/min] | 2.06 (1.02)
Stomach Mean Pressure [Mean (Standard Deviation); unit: mm Hg] | 4.44 (3.31)
Stomach High Pressure [Mean (Standard Deviation); unit: mmHg] | 313.82 (53.86)
Stomach Low pH [Mean (Standard Deviation); unit: pH] | 0 (3.84)
Stomach Median pH [Mean (Standard Deviation); unit: pH] | 2.21 (1.21)
Stomach High pH [Mean (Standard Deviation); unit: pH] | 7.48 (3.22)
Gastric Antrum Motility Index [Mean (Standard Deviation); unit: index] — Gastric antrum is the wider part of the pylorus. It resides upstream from the pyloric canal and downstream from the stomach.
  Gastric antral motility index = sum of amplitudes × number of contractions + 1.
  The average motility index in normal subjects is approximately 11. Higher values indicate either increased contractions or increased amplitudes or both. Lower values indicate either decreased contractions or decreased amplitudes or both.
  index | 17.68 (22.7)
Antrum Contractions [Mean (Standard Deviation); unit: Contractions/min] | 2.4 (2.09)
Antrum Mean Pressure [Mean (Standard Deviation); unit: mmHg] | 4.89 (3.88)
Antrum High Pressure [Mean (Standard Deviation); unit: mmHg] | 271.94 (104.4)
Antrum Low pH [Mean (Standard Deviation); unit: pH] | 0.76 (0.49)
Antrum Median pH [Mean (Standard Deviation); unit: pH] | 1.13 (0.87)
Antrum High pH [Mean (Standard Deviation); unit: pH] | 4.67 (1.81)
Duodenum Motility Index [Mean (Standard Deviation); unit: index] — Duodenal motility index = sum of amplitudes × number of contractions + 1. Higher values indicate either increased contractions or increased amplitudes or both. Lower values indicate either decreased contractions or decreased amplitudes or both.
  index | 16.84 (22.36)
Duodenum Contractions [Mean (Standard Deviation); unit: Contractions/min] | 3.13 (2.99)
Duodenum Mean Pressure [Mean (Standard Deviation); unit: mmHg] | 3.52 (1.85)
Duodenum High Pressure [Mean (Standard Deviation); unit: mmHg] | 87.07 (59.38)
Duodenum Low pH [Mean (Standard Deviation); unit: pH] | 2.33 (1.83)
Duodenum Median pH [Mean (Standard Deviation); unit: pH] | 6.30 (0.64)
Duodenum High pH [Mean (Standard Deviation); unit: pH] | 7.07 (0.60)
Small Bowel Contractions [Mean (Standard Deviation); unit: Contractions/min] | 3.88 (2.05)
Small Bowel Mean Pressure [Mean (Standard Deviation); unit: mmHg] | 4.03 (1.71)
Small Bowel High Pressure [Mean (Standard Deviation); unit: mmHg] | 143.67 (88.35)
Small Bowel Low pH [Mean (Standard Deviation); unit: pH] | 2.32 (1.87)
Small Bowel Median pH [Mean (Standard Deviation); unit: pH] | 7.36 (0.15)
Small Bowel High pH [Mean (Standard Deviation); unit: pH] | 7.89 (0.30)
Colon Contractions [Mean (Standard Deviation); unit: Contractions/min] | 2.10 (0.78)
Colon Mean Pressure [Mean (Standard Deviation); unit: mmHg] | 4.29 (1.21)
Colon High Pressure [Mean (Standard Deviation); unit: mmHg] | 177.84 (108.54)
Colon Low pH [Mean (Standard Deviation); unit: pH] | 5.19 (0.37)
Colon Median pH [Mean (Standard Deviation); unit: pH] | 6.44 (0.41)
Colon High pH [Mean (Standard Deviation); unit: pH] | 8.41 (0.38)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Lanreotide on Gastrointestinal Motility as Measured by Smart Pill
Description: If the small bowel transit time, as measured by wireless capsule endoscopy, is decreased to < 6hrs, then patient would be considered a responder and that lanreotide is efficacious.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: minutes
Arm/Group | Lanreotide
Number analyzed (Participants) | 9
minutes
  Gastric emptying time | 371.52 (45.18)
  Small bowel transit time | 392 (47.51)
  Colonic transit time | 4767 (1286)
  Small bowel and Colonic transit time | 5159 (1284)
  Whole gut transit time | 5530 (1322)
Statistical Analysis 1: Comparison: Lanreotide; Test type: Superiority; p = 0.07, t-test, 2 sided

2. Secondary Outcome: Improvement in Symptoms as Accessed by "Patient Assessment of Upper GastroIntestinal Symptom Severity Index"
Description: Improvement in symptoms assessed by improvement in Patient Assessment of Gastrointestinal Disorders Symptom Severity Index(PAGI-SYM) scores. If the PAGI-Sym scores were decreased by at least 0.7 points at 3 months when compared to baseline/pre treatment, then it will be considered that Lanreotide has significantly improved the symptom severity. Higher values represent worse symptoms.
  The participant rated each of the measured gastrointestinal symptom severity as described 0=No symptom, 1=Very Mild Symptom, 2= Mild Symptoms, 3= Moderate symptom, 4=Severe symptom, 5= Very Severe symptom.
  PAGI-SYM is a brief (20-items with 6 sub scales) symptom severity questionnaire that captures information on common upper gastrointestinal symptoms which include including Heartburn/regurgitation, Nausea/vomiting, Fullness/early satiety, bloating, Upper abdominal pain, and Lower abdominal pain. The presented data is an average of each sub scale.
Time Frame: 3 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Lanreotide
Number analyzed (Participants) | 9
score on a scale
  Heartburn/regurgitation | 1.48 (0.27)
  Nausea/vomiting | 1.00 (0.35)
  Fullness/early satiety | 2.36 (0.4)
  Bloating | 2.43 (0.47)
  Upper abdominal pain | 2.14 (0.62)
  Lower abdominal pain | 2.00 (0.51)

ADVERSE EVENTS:
Time Frame: 1 month after last dose, up to 4 months from the start for each subject.
Arm/Group | Lanreotide
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 2/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanreotide (N=9)
Difficulty swallowing wireless motility capsule pill (Investigations) | 1 (9) — One patient had difficulty in swallowing the wireless motility capsule and had a sensation that it was struck in the throat. Upon additional examination the subject was fine and was sent home.
Unable to acknowledge the passage of the wireless motility capsule through the feces (Investigations) | 1 (9) — Subject was not able to acknowledge the passage of the wireless motility capsule through the feces after the end of 4 days after ingestion. An abdominal x-ray was performed to confirm that the capsule was indeed expelled.

LIMITATIONS AND CAVEATS:
This is a pilot non-randomized study in relatively small number of subjects to identify if Lanreotide will help in alleviating the symptoms and and change gut motility in patients suffering from small bowel motility disorders. A larger study randomized study is required to confirm the findings in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-28): https://cdn.clinicaltrials.gov/large-docs/94/NCT03012594/Prot_SAP_000.pdf